CLINICAL TRIAL: NCT02325349
Title: PET/CT Molecular Imaging of Angiogenesis in Pulmonary or Head and Neck Cancers Prior to or During Chemotherapy Including Agent With Antiangiogenic Effect. A Prospective Multicentric Study of Efficacy and Tolerability.
Brief Title: PET/CT Imaging of Angiogenesis in Lung or Head and Neck Cancers Prior or During Chemotherapy With Antiangiogenic Agents
Acronym: MLAPOCHI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in protocol strategy
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P110154; 2014-000553-37 (EudraCT Number)
Record Dates: First submitted 2014-12-07; First posted 2014-12-25 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Advanced Head and Neck Carcinoma; Advanced Non-small Cell Lung Carcinoma
Keywords: Angiogenesis; Integrins; RGD PET/CT; FDG PET/CT; Predictive value; Therapeutic response; Efficacy; Tolerability
MeSH Terms: interventions — Radiopharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radiopharmaceutical (Experimental): PET/CT after intravenous administration of 2-4MBq/kg of body weight of Flotegatide (18F) or RGD (68Ga) performed prior and after 2 cycles of chemotherapy including an agent with antiangiogenic effect (two examinations in each patient)
  Interventions: Drug: radiopharmaceutical (Flotegatide (18F) or RGD (68Ga)

INTERVENTIONS:
Drug: radiopharmaceutical (Flotegatide (18F) or RGD (68Ga) — PET/CT after intravenous administration of 2-4MBq/kg of body weight of Flotegatide (18F) or RGD (68Ga) performed prior and after 2 cycles of chemotherapy including an agent with antiangiogenic effect (two examinations in each patient)

SUMMARY:
The primary objective of this Phase II study is to evaluate the use of labelled RGD ligand in PET/CT to predict and/or to early assess the efficacy of chemotherapy including an agent with antiangiogenic effect.

The predictive value of this approach will be determined by independent assessors on basis of data at the end of the treatment: RECIST 1.1 criteria for CT or MRI, PERCIST criteria for FDG PET/CT, clinical, endoscopic and histological findings.

DETAILED DESCRIPTION:
Prospective, multicentre, open label, phase II clinical trial with diagnostic radiopharmaceutical on efficacy and tolerability of 18F or 68Ga labelled RGD peptide for detection of malignant tissues expressing integrins, to predict the therapeutic response of lesions of advanced head and neck cancer or advanced non-small cells lung cancer to treatment including an agent with antiangiogenic effect.

ELIGIBILITY:
Inclusion Criteria:

* 1A. Male or female > 18year old with non-small cell lung carcinoma (NSCLC) meeting the following criteria :
* advanced NSCLC proven by histology or cytology, treatment including an agent with antiangiogenic effect scheduled
* Measurable lesions > 1 cm in short axis.
* Pretherapeutic contrast-enhanced CT of thorax and upper abdomen available for masked reading on appropriate medium
* FDG PET/CT available for masked reading on appropriate medium

  1B. Male or female > 18year old with head and neck (H&N) cancer meeting the following criteria:
* advanced H&N cancer proven by histology or cytology, treatment including an agent with antiangiogenic effect scheduled
* Measurable lesions > 1 cm in short axis.
* Pretherapeutic native and contrast enhanced CT or MRI of the head and neck available for masked reading on appropriate medium
* FDG PET/CT available for masked reading on appropriate medium
* Oto-rhino-laryngologic (ORL) examination including ORL fibroscopy and/or optionally panendoscopy.

  2. Capacity to remain without movement during the PET/CT examination 3. ECOG performance status ≤ 2 at inclusion 4. Patient with life expectancy ≥ 24 weeks after inclusion. 5. In fertile females, at inclusion the pregnancy must be ruled out 6. Volunteer and capable to follow necessary instructions during the trial 7. Informed consent signed by the patient 8. Affiliation to a social security system

Exclusion Criteria:

- 1. In patients with lung cancer: lung cancer with predominance of small-cell or pure bronchioloalveolar cancer.

2. Scheduled treatment which does not include an antiangiogenic agent 3. Patient´s physical condition not permitting participation it clinical trial according to opinion of investigator responsible of the centre 4. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Response to treatment based on RECIST criterion | Pretherapeutic Day-14, Interim Day21
  The value of pretherapeutic and interim RGD PET/CT (Pretherapeutic: D -14 to -1 before the initiation of chemotherapy with antiangiogenic agent. Interim : 21 to 1 day before the third cycle of chemotherapy with antiangiogenic agent) to early predict the therapeutic response of head and neck cancer or non-small cell lung cancer to chemotherapy with antiangiogenic agent. Final therapeutic response will be assessed at the end of the treatment, up to 24 weeks after first examination, according to criteria RECIST 1.1.
  Potential risk for the patient: two intravenous administrations of investigational product (Pretherapeutic : D -14 to -1 before the initiation of chemotherapy with antiangiogenic agent. Interim : 21 to 1 day before the third cycle of chemotherapy with antiangiogenic agent) each of them followed by PET/CT acquisition

CONTACTS AND LOCATIONS:
Overall Officials: Sona BALOGOVA, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Tenon - Assistance Publique-Hôpitaux de Paris, Paris, France